CLINICAL TRIAL: NCT04224714
Title: Clinical Study on the Correlation Between IMR（Index of Microcirculation Resistance） and FFR（Fractional Flow Reserve）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The People's Hospital of Liaoning Province (Other)
Responsible Party: Principal Investigator, Zhilin Miao, Chief physician, The People's Hospital of Liaoning Province
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTC-91616
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Myocardial Ischemia
Keywords: microcirculation resistance index (IMR); fractional flow reserve(FFR)
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Coronary heart disease patient (Experimental): Quantitative coronary angiography (QCA) showed that there was a critical lesion in the proximal or middle segment of the coronary artery (diameter stenosis rate was 50% - 70%), and the diameter of the artery was more than 2.5mm
  Interventions: Combination Product: FFR

INTERVENTIONS:
Combination Product: FFR — FFR measurement: Pressure guid wire(radianalyzer Xpress 12711) is produced in Switzerland. After the pressure of the aorta and the pressure guide wire is balanced, Send the pressure guide wire to the distal part of the lesion(more than 20 mm away from the lesion) . Adenosine is injected into the vein,then,record the FFR index 3 times and take the average value as the final measurement index.

SUMMARY:
To study the effect of myocardial microcirculation disturbance on coronary flow reserve fraction, compare the evaluation value of IMR, FFR and QCA on myocardial ischemia, and discuss the correlation among them.

DETAILED DESCRIPTION:
In this study, 60 patients with critical lesions indicated by coronary angiography will be admitted. The investigators collected the basic clinical data (gender, age, body mass index, smoking history, hypertension, diabetes, hyperlipidemia), laboratory data (creatinine, cholesterol, triglycerides) and measured their FFR and IMR.

ELIGIBILITY:
Inclusion Criteria:(1) Age: 18-75 years old, unlimited for men and women;

(2) Quantitative coronary angiography (QCA) showed that there was a critical lesion in the proximal or middle segment of the coronary artery (diameter stenosis rate was 50% - 70%), and the diameter of the artery was more than 2.5mm;

(3) Agree to participate in the study and sign informed consent

-

Exclusion Criteria:(1) Patients with acute myocardial infarction within one month;

(2) Patients with congenital heart disease, severe valve disease, dilated cardiomyopathy, pulmonary heart disease and hypertrophic cardiomyopathy;

(3) With severe heart failure (NYHA cardiac function grade ≥ grade III or left ventricular ejection fraction < 35%);

(4) Patients with less than 1 year of stent implantation or with coronary artery bypass grafting;

(5) Patients with left main lesion, severe distorted calcification, open lesion, bifurcated lesion or complete occlusion;

(6) Patients with severe hepatorenal insufficiency;

(7) Contraindications to adenosine, aspirin and clopidogrel;

(8) Patients with advanced tumor or life expectancy less than 1 year;

(9) Patients with severe asthma or uncontrolled asthma;

(10) Women in pregnancy.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
IMR | one hour
  Resistance index of microcirculation

CONTACTS AND LOCATIONS:
Locations (1):
- The people's hospital of LiaoNing Province, Shenyang, Liaoning, China